CLINICAL TRIAL: NCT04629027
Title: Establishment of a Comprehensive Evaluation System for the Efficacy of Immunologic Checkpoint Inhibitors in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Evaluation System for the Efficacy of Immunologic Checkpoint Inhibitors in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jian Fang, Principal Investigator, Peking University Cancer Hospital & Institute
Other Study IDs: 2020-2-2153
Record Dates: First submitted 2020-11-06; First posted 2020-11-16 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: advanced lung cancer; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — the patients receive necessary treatment without special intervention

SUMMARY:
Inhibitors of programmed cell death protein 1 (PD-1) and programmed cell death ligand 1 (PD-L1) are effective therapies for metastatic NSCLC lacking sensitizing EGFR or ALK mutations. First-line combination regimens that include a PD-1 or PD-L1 inhibitor may maximize the chance of response and lead to prolonged survival. PD-L1 expression is the only validated predictive biomarker for selecting pembrolizumab treatment. However, it is far from being the ideal biomarker and its role in predicting efficacy from ICPIs remains undefined due to conflicting results from randomized clinical trials. The selection of patients most likely to benefit from immunotherapy is crucial in order to avoid exposure to potentially toxic and ineffective drugs as well as to prevent inappropriate allocation of health resources. Further studies are clearly needed to better understand the mechanism of action of immunotherapy in vivo thus allowing the identification of other predictive biomarkers. Therefore, our research team intends to explore advanced non-small cell lung cancer treated with immune checkpoint inhibitors, by combining the evaluation criteria of solid tumor efficacy evaluation criteria (RECIST1.1), clinical pathological characteristics of patients, and dynamic monitoring of peripheral blood molecular biological markers, finding the correlation with the efficacy of immunotherapy, establish a detection mode for selecting patients with clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

Ages ≥18 years of age. Histologically confirmed stage IIIB-IV non-squamous non-small cell lung cancer. Life expectancy of at least 3 months.

Exclusion Criteria:

* Previous treatment . Untreated CNS metastases. Active autoimmune disease. Surgery or significant traumatic injury. Active infection. History of allergy or hypersensitivity to immunotherapy components. Women are breastfeeding or pregnant. Requiring systemic treatment with either corticosteroids or other immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients can accepted immune checkpoint inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
circulating tumor cell | 3 year
  The selection of patients most likely to benefit from immunotherapy is crucial in order to avoid exposure to potentially toxic and ineffective drugs.
T cell marker | 3 year
  The selection of patients most likely to benefit from immunotherapy is crucial in order to avoid exposure to potentially toxic and ineffective drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Fang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China